CLINICAL TRIAL: NCT01003522
Title: Randomised Evaluation of Stents to Open Restricted Airways in Patients With Centrally Placed Non-small Cell Lung Cancer (RESTORE-AIR)
Brief Title: Evaluation of Stents to Open Restricted Airways in Patients With Centrally Placed Non-small Cell Lung Cancer
Acronym: RESTORE-AIR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Dr Mary O'Brien, Royal Marsden NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR2987
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Bronchial stents; Airway obstruction; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Airway Obstruction | interventions — Blood Specimen Collection; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm A (Other): Stenting of central lesion and subsequent standard palliative treatment and dyspnoea symptom control
  Interventions: Other: Arterial puncture; Other: Venepuncture; Procedure: General anaesthetic; Procedure: Inpatient stays; Other: Walking test; Other: Spirometry & flow volume loop assessment; Other: Biopsy material
- Treatment Arm B (Other): Standard palliative treatment and standard dyspnoea symptom control.
  Interventions: Other: Arterial puncture; Other: Venepuncture; Other: Walking test; Other: Spirometry & flow volume loop assessment

INTERVENTIONS:
Other: Arterial puncture — Patients will undergo arterial blood gas sampling from the radial artery. This will be done by experienced doctors who are highly skilled in this procedure.
Other: Venepuncture — Blood samples for baseline biochemistry, full blood count, and clotting screen will be taken. In patients additionally providing optional consent blood will be taken for laboratory based basic science research into lung cancer carcinogenesis and pharmacogenetics. Blood will be taken by qualified and experienced nurses, doctors and phlebotomists.
Procedure: General anaesthetic — Patients randomised into the stenting arm will undergo rigid bronchoscopy under general anaesthetic.
  Arms: Treatment Arm A
Procedure: Inpatient stays — Patients randomised into the stenting arm will be admitted overnight for the procedure
  Arms: Treatment Arm A
Other: Walking test — All patients will be asked to complete a 6 minute walking test at baseline and on day 15. Patients randomised into the stent arm (Arm A) will complete a further 6 minute walking test at 24 hours post-stent
Other: Spirometry & flow volume loop assessment — All patients will undergo spirometry and flow volume loop assessments at baseline and on day 15.
Other: Biopsy material — For patients randomised to stenting and giving additional voluntary consent, 2 pairs of biopsies of tumour tissue, and 1 pair of biopsies of normal airways tissue will be taken for basic scientific research into lung cancer carcinogenesis, and pharmacogenetics.
  Arms: Treatment Arm A

SUMMARY:
To investigate whether the use of airways stents (metal tubes to open and keep open narrowed airways) together with the standard treatment increases the proportion of patients who can complete a 6min walking distance (6MWD) test at 2 weeks +/- 2days in patients with breathlessness due to lung cancer, when compared to standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed written consent in the English language
* Able and willing to attend St Georges Hospital / Royal Marsden Hospital for stent insertion (if allocated) and documentation of 6 minute walking distance.
* Willing to re-attend for follow-up and 6 minute walking distance at St Georges Hospital / Royal Marsden Hospital 2 weeks later (all patients)
* Diagnosis of non-small cell lung cancer with centrally placed tumour with some degree of airway obstruction from information from bronchoscopy or CT scan.
* ECOG Performance status: 0-3

Exclusion Criteria:

* Relative contraindications to stenting, e.g. bleeding abnormality or anticoagulation problems.
* Pregnancy
* Radically treatable disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is the proportion of patients achieving a 50% improvement in the distance walked after 2 weeks +/- 2 days of treatment as compared to their pre-treatment assessment.

SECONDARY OUTCOMES:
To compare arterial blood gases (oxygenation of blood) from baseline to 2 weeks +/- 2 days in the stented group, compared with the standard treatment group.
To compare lung function tests from baseline to 2 weeks +/- 2 days in the stented group, compared with the standard treatment group.
To compare other symptoms such as anxiety and breathlessness, as measured by standard scales (e.g. VAS, Borg scales) from baseline to 2 weeks +/- 2 days in the stented group, compared with the standard treatment group
To measure quality of life with standard questionnaires
To compare survival rates at 6 months and 1 year between the stented group and standard treatment group
To document any subsequent treatments given to patients in each group
To establish the feasibility of collecting fresh and formalin fixed, paraffin embedded tumour and normal bronchial tissue, and germ-line DNA for future research into NSCLC carcinogenesis and corollary translational work
Formal objective response assessment is not required at 3 months, but where this is possible, this will be described

CONTACTS AND LOCATIONS:
Overall Officials: Mary O'Brien, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom